CLINICAL TRIAL: NCT01129700
Title: Short-course Preoperative Chemoradiotherapy Followed by Delayed Operation for Locally Advanced Rectal Cancer: Phase II Multi-institutional Study
Brief Title: Short-course Preoperative Chemoradiotherapy Followed by Delayed Operation for Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, DAE YONG KIM, Principal Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-10-458
Record Dates: First submitted 2010-05-13; First posted 2010-05-25 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Rectal Cancer
Keywords: rectal cancer, short-course, chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- short-course CRT-5FU (Experimental)
  Interventions: Radiation: Radiation: short-course preoperative chemoradiotherapy

INTERVENTIONS:
Radiation: Radiation: short-course preoperative chemoradiotherapy — Drug: 5-Fluorouracil 5-Fluorouracil is administered intravenously at a dose of 400 mg/m2 once daily continuous regimen during RT(5 days).
  Radiation: Localization, simulation and immobilization Radiation dose and planning Total dose 25Gy, 5 fractions (5 Gy/day).

SUMMARY:
Concurrent chemoradiotherapy (CRT)

* Radiotherapy 25 ㏉/5 fractions (start concomitantly at D1)

  * ↓ ↓ ↓ ↓ ↓

    * Radical surgery 6 weeks after completion of chemoradiotherapy

      * ↑ ↑ ↑ ↑ ↑ D1 - - - - - D5
* 5-Fluorouracil 400㎎/㎡/day + LV 20㎎/㎡/day IV bolus during the radiotherapy

DETAILED DESCRIPTION:
Radiotherapy using tomotherapy is delivered in 5 Gy daily fractions for a total of 25 Gy in 5 fractions.

A bolus injection of 5-fluorouracil (400 mg/m2/d)and leucovorin (20 mg/m2/d) is delivered concurrently on day 1-5 during radiotherapy.

Total mesorectal excision is performed within 6±2 weeks. The pathological response of downstaing is the study endpoint.

ELIGIBILITY:
Inclusion Criteria :

* Pathologically proven diagnosis of adenocarcinoma of the rectum (located within 8㎝ above the anal verge)
* Locally advanced and curatively resectable tumor(cT3-4 classification) evaluated with magnetic resonance imaging(MRI) with or without transrectal ultrasonography(TRUS)
* Age ≥18
* Performance Status(ECOG) 0-2
* CBC/differential obtained within 14 days prior to registration on study, with adequate bone marrow function defined as follows: Hemoglobin ≥ 10 g/dl, Absolute neutrophil count(ANC) ≥ 1,500 cells/㎣, Platelets ≥ 100,000cells/㎣
* Metabolic panel within 14 days prior to registration on study, with adequate liver and renal function defined as follows: AST and ALT ≤ 60 IU/L, bilirubin ≤ 1.5 mg/dl, serum creatinine ≤ 1.5 mg/dl
* Patient must provide study-specific informed consent prior to study entry

Exclusion Criteria :

* Any evidence of distant metastases(M1)
* Prior invasive malignancy (except non-melanomatous skin cancer and uterine cervical cancer in situ) unless disease free to a minimum of 3 years
* Hereditary rectal cancer; Familial adenomatous polyposis(FAP), Hereditary non-polyposis colorectal cancer(HNPCC), etc.
* Impending obstruction (except the case with colostomy)
* Severe, active comorbidity inappropriate to CRT as follows; Acute bacterial or fungal infection, transmural myocardial infarction within the last 6 months, unstable arrhythmia, angina and/or congestive heart failure, unstable arrhythmia
* Pregnancy or women of childbearing potential who are sexually active and not willing/able to use medically acceptable forms of contraception
* Unresected synchronous colon carcinoma
* Clinically unresectable rectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the pathologic response | After surgery with pathology data
  downstaging(ypT0-2N0M0)rate

SECONDARY OUTCOMES:
Tumor regression grade & MR volumetry | After surgery with pathology data for TRG, at the pretreatment work-up and 1-4 days befor surgery
  To evaluate the tumor regression grade & MR volumetry
Acute/ late toxicities | preoperative CCRT to 3 months after surgery
  To evaluate the acute and late toxicities

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea